CLINICAL TRIAL: NCT03279237
Title: A Pilot Study of FOLFIRINOX in Combination With Neoadjuvant Radiation for Gastric and GE Junction Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jennifer Wo, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-311; U19CA021239-37 (NIH)
Record Dates: First submitted 2017-09-07; First posted 2017-09-12 (Actual); Results first posted 2020-05-07 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: GastroEsophageal Cancer
Keywords: GastroEsophageal Cancer
MeSH Terms: interventions — Irinotecan; Oxaliplatin; Leucovorin; Fluorouracil; Paclitaxel; Albumin-Bound Paclitaxel; Radiotherapy; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- FOLFIRINOX + pre-operative radiation (Experimental): * FOLFIRINOX is a combination of 4 drugs that is administered twice per cycle
    * Oxaliplatin is administered intravenously
    * Leucovorin is administered intravenously
    * Irinotecan is administered intravenously
    * 5-Fluorouracil is administered intravenously
  * Paclitaxel and Carboplatin will be given concurrently with radiation therapy every 7 days
  Interventions: Drug: Irinotecan; Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5-Fluorouracil; Drug: Paclitaxel; Radiation: Radiation Therapy; Drug: Carboplatin

INTERVENTIONS:
Drug: Irinotecan — May help shrink tumor before surgery.
  Other Names: Camptosar
Drug: Oxaliplatin — May help shrink tumor before surgery.
  Other Names: Eloxatin
Drug: Leucovorin — May help shrink tumor before surgery.
Drug: 5-Fluorouracil — May help shrink tumor before surgery.
  Other Names: Efudex
Drug: Paclitaxel — Paclitaxel may stop cancer cells from growing and spreading.
  Other Names: Abraxane
Radiation: Radiation Therapy — May help shrink tumor.
Drug: Carboplatin — Carboplatin may stop cancer cells from growing.

SUMMARY:
This research study is studying a combination of interventions as a possible treatment for gastroesophageal (GE) junction cancer.

The interventions involved in this study are:

-FOLFIRINOX which is made up of 4 different drugs:

* 5-Fluorouracil (5-FU)
* Oxaliplatin
* Irinotecan
* Leucovorin
* Paclitaxel
* Carboplatin
* Proton Beam Radiation Therapy

DETAILED DESCRIPTION:
This research study is a Pilot Study, which is the first time investigators are examining this study intervention.

In this research study, the investigators are studying the combination of FOLFIRINOX followed by radiation with paclitaxel and carboplatin before surgery. The investigators believe that this intervention may help decrease the growth and spread of the cancer cells.

FOLFIRINOX has shown to be very effective in patients whom disease has spread. The investigators are evaluating this regimen to see if there is an increase in curability when the cancer has not spread.

The FDA (the U.S. Food and Drug Administration) has approved FOLFIRINOX as a treatment option for this disease.

The FDA has not approved Paclitaxel or Carboplatin for this specific disease but they have both been approved for other uses.

FOLFIRINOX is a combination of 4 chemotherapy agents that may help shrink the tumor before surgery.

Carboplatin may stop the cancer cells from growing and paclitaxel may stop the cancer cells from growing and spreading

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed T 3/4 or N+ (> 1 cm in size or FDG avid) gastric or gastroesophageal (GE) junction cancer. Diagnosis must be confirmed by the Mass General Hospital pathology department.
* Age 18 years or older. There will be no upper age restriction.
* ECOG performance status ≤ 1
* Life expectancy of greater than 3 months
* Participants must have adequate organ and marrow function as defined below:

  * absolute neutrophil count ≥ 1,500 cells/mm3
  * platelets ≥ 75,000 cells/mm3
  * total bilirubin ≤ 1.5 x upper limit of normal, or, for patients who have
  * undergone biliary stenting, total bilirubin of ≤ 2 or two down trending values.
  * AST(SGOT) ≤ 2.5 × upper limit of normal
  * ALT (SGPT) ≤ 2.5 x upper limit of normal
  * creatinine ≤ 1.5 mg/dL, or
  * creatinine clearance ≥ 30 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
* The effects of both radiation therapy and the chemotherapy agents used in this trial are known to be teratogenic. Therefore, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation plus 30 days from the last date of study drug administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Evidence of metastatic disease as determined by chest CT scan, abdomen/pelvis CT scan (or MRI with gadolinium and/or manganese) within six weeks of study entry. Distant nodal disease is allowed if it is in the radiation port.
* Any prior chemotherapy, targeted/biologic therapy, or radiation for treatment of the participant's gastric or GE junction cancer.
* Receipt of chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Treatment of other invasive carcinomas within the last five years with greater than 5% risk of recurrence at time of eligibility screening. Carcinoma in-situ and basal cell carcinoma/ squamous cell carcinoma of the skin are allowed.
* Receipt of any other investigational agents within 4 weeks preceding the start of study treatment.
* Serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator), such as significant cardiac or pulmonary morbidity (e.g. congestive heart failure, symptomatic coronary artery disease and/or cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months, or ongoing infection as manifested by fever.
* History of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance or drug intake.
* Pregnant women are excluded from this study because radiation therapy and the chemotherapy agents to be used have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued while the mother is receiving protocol therapy.
* Major surgery, excluding laparoscopy, within 4 weeks of the start of study treatment, without complete recovery.
* No concurrent administration of cimetidine (as it can decrease the clearance of 5-FU). Another H2-blocker or proton pump inhibitor may be substituted before study entry.
* Known, existing uncontrolled coagulopathy.
* Prior systemic fluoropyrimidine therapy (unless given in an adjuvant setting and at least six months earlier). Prior topical fluoropyrimidine use is allowed.
* Known hypersensitivity to 5-fluorouracil or known DPD deficiency.
* History of allergic reaction(s) attributed to compounds of similar chemical or biologic composition to 5-fluorouracil, irinotecan, or oxaliplatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2024-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Wo, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wo JY, Clark JW, Eyler CE, Mino-Kenudson M, Klempner SJ, Allen JN, Keane FK, Parikh AR, Roeland E, Drapek LC, Ryan DP, Corcoran RB, Van Seventer E, Fetter IJ, Shahzade HA, Khandekar MJ, Lanuti M, Morse CR, Heist RS, Ulysse CA, Christopher B, Baglini C, Yeap BY, Mullen JT, Hong TS. Results and Molecular Correlates from a Pilot Study of Neoadjuvant Induction FOLFIRINOX Followed by Chemoradiation and Surgery for Gastroesophageal Adenocarcinomas. Clin Cancer Res. 2021 Dec 1;27(23):6343-6353. doi: 10.1158/1078-0432.CCR-21-0331. Epub 2021 Jul 30. PMID 34330715

RESULTS

PARTICIPANT FLOW:
Groups:
- FOLFIRINOX + pre-operative radiation: * FOLFIRINOX is a combination of 4 drugs that is administered twice per cycle
    * Oxaliplatin is administered intravenously
    * Leucovorin is administered intravenously
    * Irinotecan is administered intravenously
    * 5-Fluorouracil is administered intravenously
  * Paclitaxel and Carboplatin will be given concurrently with radiation therapy every 7 days
  Irinotecan: May help shrink tumor before surgery.
  Oxaliplatin: May help shrink tumor before surgery.
  Leucovorin: May help shrink tumor before surgery.
  5-Fluorouracil: May help shrink tumor before surgery.
  Paclitaxel: Paclitaxel may stop cancer cells from growing and spreading.
  Radiation Therapy: May help shrink tumor.
  Carboplatin: Carboplatin may stop cancer cells from growing.
Period: Overall Study
Arm/Group | FOLFIRINOX + pre-operative radiation
Started | 25
Chemo-radiation | 23
Surgical Resection | 20
Completed | 20
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | FOLFIRINOX + Pre-operative Radiation
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 60 [30 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: The Completion Rate of Chemotherapy in Combination With Chemoradiation
Description: The number of participants that complete the assigned study intervention.
Time Frame: 21 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | FOLFIRINOX + pre-operative radiation
Number analyzed (Participants) | 25
Participants | 23

2. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: The number of participants that experienced at least one treatment related adverse event as assessed by Common Terminology Criteria for Adverse Events (CTCAE v4.0).
Time Frame: From the start of treatment until 30 days after the end of treatment (up to approximately 25 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | FOLFIRINOX + pre-operative radiation
Number analyzed (Participants) | 25
Participants | 25

3. Secondary Outcome: Clinical Response Rate
Description: The number of participants that achieved a clinical response following treatment. Clinical response is defined as achieving a best overall response of a complete response (CR) or a partial response (PR).
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: After 4 and 8 cycles of FOLFIRINOX (8 and 16 weeks); and 3-4 weeks after chemo radiation (24-25 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | FOLFIRINOX + pre-operative radiation
Number analyzed (Participants) | 25
Participants | 20

4. Secondary Outcome: Pathologic Complete Response Rate
Description: The number of participants that achieve a pathologic complete response at surgery following FOLFIRINOX and chemoradiation. All patients will undergo a full pathological review of their surgical specimen according to the American Joint Committee on Cancer (AJCC) Staging Classification, 6th edition. Initial gross evaluation and identification of resection margins will be performed jointly by the surgeon and the pathologist. Pathological complete response will be defined as the absence of any viable tumor cells within the pathologic specimen.
Time Frame: 29 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | FOLFIRINOX + pre-operative radiation
Number analyzed (Participants) | 25
Participants | 7

5. Secondary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) is defined as the time from the date of first dosing to the first documentation of radiographic disease progression per Response Evaluation Criteria In Solid Tumors (RECIST v1.1) or death due to any cause, whichever occurs first. Subjects who are alive with no documented progressive disease by the data cutoff date for PFS analysis will be censored at the date of their last evaluable disease assessment.
  Progressive Disease (PD) is defined as having at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: 5 Years
Reporting Status: Not Posted

6. Secondary Outcome: Overall Survival
Description: The number of participants alive five years after the start of treatment. Overall survival (OS) is measured as the time from the date of first dosing until death due to any cause. If there is no death reported for a subject by the data cut-off date for overall survival analysis, OS will be censored at the last known alive date.
Time Frame: 5 Years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the start of treatment until 30 days after the end of treatment (up to approximately 25 weeks)
Description: Serious adverse events were defined as grade 3 or greater adverse events that were deemed to be at least possibly, probably, or definitely related to treatment. Non-serious adverse events were not captured.
Arm/Group | FOLFIRINOX + pre-operative radiation
All-Cause Mortality (participants affected / at risk) | 1/25
Serious Adverse Events (participants affected / at risk) | 24/25
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFIRINOX + pre-operative radiation (N=25)
Lymphopenia/Leukopenia/Neutropenia (Blood and lymphatic system disorders) | 21
Febrile Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Anemia (Blood and lymphatic system disorders) | 3
Hypokalemia/Hyponatremia/Hypocalcemia (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 2
Weight loss (Metabolism and nutrition disorders) | 1
Nausea/vomiting (Metabolism and nutrition disorders) | 4
Diarrhea (Metabolism and nutrition disorders) | 4
Dysphagia (Metabolism and nutrition disorders) | 1
Mucositis, Oral (Metabolism and nutrition disorders) | 1
Gastrointestinal, Other (Metabolism and nutrition disorders) | 1
Infection (Metabolism and nutrition disorders) | 2
Hypotension (Metabolism and nutrition disorders) | 2
Fatigue (Metabolism and nutrition disorders) | 1
ALT/ALK phosphatase elevated (Metabolism and nutrition disorders) | 1
Cardiac (Metabolism and nutrition disorders) | 1
Acute kidney injury (Metabolism and nutrition disorders) | 1
Aspiration (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-14): https://cdn.clinicaltrials.gov/large-docs/37/NCT03279237/Prot_SAP_000.pdf